CLINICAL TRIAL: NCT02588053
Title: Does Long-Term Natalizumab (NTZ) Therapy Normalize Brain Atrophy Rates and Quality of Life (QOL) in Relapsing Remitting Multiple Sclerosis (RRMS)? A Longitudinal Study Using Whole Brain, Neocortical and Subcortical Atrophy Rates and Patient Reported Outcomes (PROs).
Brief Title: Does Long-Term Natalizumab (NTZ) Therapy Normalize Brain Atrophy Rates and Quality of Life (QOL) in Relapsing Remitting Multiple Sclerosis (RRMS)?
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 13-2927; UL1TR001082 (NIH)
Record Dates: First submitted 2014-07-16; First posted 2015-10-27 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Aims: To determine how effective long term Natalizumab (NTZ) therapy is in slowing the progression of whole brain atrophy. Whole brain atrophy rates will be measured through magnetic resonance imaging (MRI) scans and compared between patients with Multiple Sclerosis (MS) who have been using NTZ for at least 2 years versus age and gender-matched healthy controls. The primary outcome will be whole brain atrophy rate measured as the percent change in brain volume (PBVC) over a two-year period.

Primary hypothesis:

The investigators hypothesize that long term (>2 years) NTZ therapy will slow the rate of whole brain atrophy in patients with Multiple Sclerosis (MS) (as measured by percent change in brain volume), reaching a whole brain atrophy rate similar to that of non-MS controls (a true "disease activity free" state).

ELIGIBILITY:
Inclusion Criteria:

* 18-55 inclusive years of age at the time of informed consent
* Diagnosis of relapsing multiple sclerosis as defined by the 2010 revised McDonald criteria
* Currently taking Tysabri

Exclusion Criteria:

* Systemic steroid users
* comorbidities that could confound MRI outcomes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Relapsing Multiple Sclerosis and Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in Brain Atrophy Rate | Baseline, Year 1, and Year 2

SECONDARY OUTCOMES:
Change in Mean Cortical Thickness | Baseline, Year 1, and Year 2
Change in Neocortical Gray Matter Volume | Baseline, Year 1, and Year 2
Change in Subcortical Gray Matter Volume | Baseline, Year 1, and Year 2

OTHER OUTCOMES:
Change in Patient-reported Quality of Life | Baseline, Year 1, and Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Miravalle, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States